CLINICAL TRIAL: NCT00971906
Title: A Randomized, Single-blind, Dose-Ranging, Study to Evaluate Immunogenicity, Safety and Tolerability of Different Formulations of Adjuvanted and Non Adjuvanted Egg-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Subjects 18 or More Years of Age
Brief Title: Immunogenicity, Safety and Tolerability of Two Doses of Adjuvanted and Non-adjuvanted Swine Origin A/H1N1 Monovalent Influenza Vaccine in Healthy Subjects 18 or More Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V111_02; 2009-013671-21 (EudraCT Number)
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2011-10

CONDITIONS: Pandemic Influenza
Keywords: Pandemic influenza; Vaccine

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- low dose of antigen + low dose of adjuvant (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- high dose of antigen + high dose of adjuvant (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- high dose of antigen (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine

INTERVENTIONS:
Biological: Monovalent A/H1N1 influenza vaccine — This trial will be performed at multiple study sites in a population of healthy adults and elderly. Subjects will be randomized to receive two IM injections of low dose of antigen & adjuvant,or high dose of antigen & adjuvant, or high dose of antigen, according to the study groups

SUMMARY:
This present study, randomized, single-blind, dose-ranging, multicenter study, will evaluate immunogenicity, safety and tolerability of two doses of an adjuvanted and not-adjuvanted new swine-origin influenza A/H1N1 virus monovalent subunit vaccine in healthy adult and elderly subjects. A booster dose will be administered 12 months after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and above on the day of enrollment;
2. Individuals in good health
3. Individuals are able to comply with all study procedures
4. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Individual not able to comprehend and to follow all required study procedures;
2. History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
3. Any serious chronic or progressive disease according to judgment of the investigator
4. History of any anaphylaxis, serious vaccine reactions, to any excipients.
5. Adjuvanted influenza vaccine or documented confirmed or suspected influenza disease within 3 months prior to Day 1;
6. Receipt of another investigational agent within 4 weeks prior to enrollment, or before completion of the safety follow-up period in this or in another study; unwilling to refuse participation in another clinical study through the end of this study;
7. Any other vaccines within 4 weeks prior to enrollment or who are planning to receive any vaccine within 4 weeks from the study vaccines; only exception being plain seasonal influenza vaccines which are allowed until 1 week prior to and after 1 week study vaccinations.
8. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks;
9. Axillary temperature ≥ 38°C or oral temperature ≥ 38.5°C within 3 days of intended study vaccination;
10. Known or suspected impairment/alteration of immune function, for example resulting from a receipt of immunosuppressive therapy within 60 days prior to Visit 1;
11. History of progressive or severe neurological disorders;
12. Surgery planned during the study period that in the Investigator's opinion would interfere with the study visits schedule;
13. Female of childbearing potential, not used any acceptable contraceptive methods for at least 2 months prior to study entry;
14. Female pregnant or nursing (breastfeeding) mothers or females of childbearing potential do not plan to use acceptable birth control measures during the first 3 weeks after vaccination;
15. Members of the research staff or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To identify the preferred vaccine formulation, dosage (antigen & adjuvant), schedule (one or two administrations) of the H1N1 sw monovalent vaccine in adults | 43 days after first vaccination

SECONDARY OUTCOMES:
To evaluate immunogenicity against A/California H1N1sw strain after booster dose of egg-derived seasonal trivalent, MF59 adjuvanted vaccine Fluad, recommended for 2010/2011 season, administered 12 months after primary course according to CHMP criteria | 3 weeks after booster vaccination

CONTACTS AND LOCATIONS:
Locations (4):
- Gent, Antwerpen, Antwerp, Belgium
- Munchen, Wurzburg, Balve, Leipzig, Magdeburg, Hamburg, Rostock, Mainz, Mainz, Germany
- Switzerland (2):
  - Basel
  - Zurich

REFERENCES:
- [Derived] Hatz C, von Sonnenburg F, Casula D, Lattanzi M, Leroux-Roels G. A randomized clinical trial to identify the optimal antigen and MF59((R)) adjuvant dose of a monovalent A/H1N1 pandemic influenza vaccine in healthy adult and elderly subjects. Vaccine. 2012 May 14;30(23):3470-7. doi: 10.1016/j.vaccine.2012.03.017. Epub 2012 Mar 22. PMID 22446638